CLINICAL TRIAL: NCT00422669
Title: Optimize RV Selective Site Pacing Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment significantly below protocol expectations
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 604
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Cardiac Pacing, Artificial; Cardiac Pacemaker, Artificial
Keywords: Pacemaker; Implantable Pulse Generator (IPG); AV Conduction Disturbance; Select Site Pacing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RV Mid-Septal Pacing (Active Comparator): Pacing lead is placed in the right ventricle at the middle of the muscle separating the right and left sides of the heart
  Interventions: Device: Medtronic Dual-Chamber Pacemaker; Device: Medtronic SelectSecure 3830 Lead
- RV Apical Pacing (Active Comparator): Pacing lead is placed at the bottom of the right ventricle of the heart, in the right ventricular apex
  Interventions: Device: Medtronic Dual-Chamber Pacemaker; Device: Medtronic SelectSecure 3830 Lead

INTERVENTIONS:
Device: Medtronic Dual-Chamber Pacemaker — A Medtronic market-approved dual-chamber implantable pulse generator (IPG)
Device: Medtronic SelectSecure 3830 Lead — Medtronic market-approved SelectSecure Model 3830 bipolar pacing lead

SUMMARY:
The purpose of the Optimize RV study is to determine the long-term effect of selective site pacing. Selective site pacing refers to which area of the right ventricle the lead is placed. The goal of select site pacing is to improve how the heart contracts when paced in the ventricle. By pacing in select sites, it is possible to better copy the natural pattern of contraction of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are expected to be paced in the right ventricle (RV) greater than 90 percent of the time
* Subjects with an ejection fraction of greater than 40 percent within 3 months prior to enrollment
* Subjects greater than 18 yrs of age
* Subjects that are indicated for a dual chamber pacemaker
* Subjects that will be implanted with a market released dual chamber Medtronic pacemaker and 3830 SelectSecure Lead in the ventricle

Exclusion Criteria:

* Subjects indicated for cardiac resynchronization therapy (CRT) device (based on American College of Cardiology/American Heart Association/Heart Rhythm Society guidelines)
* Subjects indicated for an implantable cardiac defibrillator (ICD)
* Subjects with permanent atrial fibrillation (AF)
* Subjects with expected managed ventricular pacing turned on
* Subjects with a previously implanted pacemaker, ICD, or CRT device
* Subjects with an myocardial infarction (MI) within 3 months prior to enrollment
* Subjects that received bypass surgery within 3 months prior to enrollment
* Subjects that had valve replacement within 3 months prior to enrollment
* Subjects where a RV lead cannot be placed, (i.e., complex congenital heart disease
* Subjects with a mechanical right heart valve
* Women who are pregnant or nursing
* Significant co-morbidity preventing study completion
* Terminal conditions with a life expectancy of less than two years
* Participation in another study that would confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Optimize RV Team, Study Chair — Medtronic
Locations (22):
- United States (16):
  - Bridgeport, Connecticut
  - Clearwater, Florida
  - Hudson, Florida
  - Des Moines, Iowa
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Southfield, Michigan
  - Saint Paul, Minnesota
  - Omaha, Nebraska
  - Cleveland, Ohio
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
- Montreal, Canada
- Hong Kong, China
- Ramat Gan, Israel
- Italy (2):
  - Florence
  - Rovigo
- Doha, Qatar

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollments in the Optimize RV trial began in March of 2007. The study was terminated early on March 26, 2009 after 205 subjects had been enrolled.
Pre-assignment Details: Seven subjects did not meet inclusion/exclusion criteria.
Groups:
- Not Randomized: 7 of the 205 subjects did not meet inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | RV Mid-Septal Pacing | RV Apical Pacing | Not Randomized
Started | 98 (Data required for analysis was not collected due to early termination. Analysis will not be done.) | 100 (Data required for analysis was not collected due to early termination. Analysis will not be done.) | 7
Completed | 0 (Data required for analysis was not collected due to early termination. Analysis will not be done.) | 0 (Data required for analysis was not collected due to early termination. Analysis will not be done.) | 0
Not Completed | 98 | 100 | 7
Not completed — The study was terminated early. | 98 | 100 | 7

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: 7 of the 205 subjects did not meet in/exclusion criteria so they were not randomized.
- Total: Total of all reporting groups
Arm/Group | RV Mid-Septal Pacing | RV Apical Pacing | Not Randomized | Total
Number analyzed (Participants) | 98 | 100 | 7 | 205
Age Continuous [Mean (Standard Deviation); unit: years] | 77.1 (11.2) | 77.1 (10.5) | NA (NA) — The data were not submitted due to not meeting in/exclusion criteria | 77.1 (10.8)
Gender [Number; unit: participants]
  Female | 37 | 39 | NA — The data were not submitted due to not meeting in/exclusion criteria | 76
  Male | 61 | 61 | NA — The data were not submitted due to not meeting in/exclusion criteria | 122
Region of Enrollment [Number; unit: participants]
  United States | 75 | 78 | 7 | 160
  Canada | 5 | 6 | 0 | 11
  Israel | 5 | 4 | 0 | 9
  Italy | 13 | 12 | 0 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Change in Left Ventricular (LV) Ejection Fraction From Baseline to Two Year Follow-up
Description: Left ventricular ejection fraction (LVEF) will be measured at baseline and two year follow-up for the group of pacing at RV Mid-Septum and the group of pacing at Apex. The change in LVEF from baseline to two year follow-up will be compared between two groups to identify if pacing at selective RV sites (Mid-Septum or Apex) will have a different long term impact on the change in LVEF.
Time Frame: Baseline and 24 months
Population: Data required for the analysis were not collected due to early study termination. Analysis will not be done.
Arm/Group | RV Mid-Septal Pacing | RV Apical Pacing | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: The Change in LVEF From Two Week Visit to Two Year Follow-up
Description: Left ventricular ejection fraction (LVEF) will be measured at two week visit and 2 year follow-up for the group of pacing at RV Mid-Septum and the group of pacing at Apex. The change in LVEF from two week visit to 2 year follow-up will be compared between two groups to identify if pacing at selective RV sites (Mid-Septum or Apex) will have a different long term impact on the change in LVEF.
Time Frame: Baseline and 24 months
Population: Data required for the analysis were not collected due to early study termination. Analysis will not be done.
Arm/Group | RV Mid-Septal Pacing | RV Apical Pacing | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: The Change in Six-minute Hall Walk Distance
Description: The change in six-minute hall walk distance will be measured at two week visit and 2 year follow-up for the group of pacing at RV Mid-Septum and the group of pacing at Apex. The change in six-minute hall walk distance will be compared between two groups to identify if pacing at selective RV sites (Mid-Septum or Apex) will have a different long term impact on the change in six-minute hall walk distance.
Time Frame: Baseline and 24 months
Population: Data required for the analysis were not collected due to early study termination. Analysis will not be done.
Arm/Group | RV Mid-Septal Pacing | RV Apical Pacing | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: The Change in Left Ventricular (LV) End Systolic Volume (Diastolic Volume) After Two Years Follow-up
Description: LV end systolic volume (diastolic volume)will be measured at baseline and 2 year follow-up for the group of pacing at RV Mid-Septum and the group of pacing at Apex. The change in LV end systolic volume (diastolic volume)from two week visit to 2 year follow-up will be compared between two groups to identify if pacing at selective RV sites (Mid-Septum or Apex) will have a different long term impact on the change in LV end systolic volume (diastolic volume).
Time Frame: Baseline and 24 months
Population: Data required for the analysis were not collected due to early study termination. Analysis will not be done.
Arm/Group | RV Mid-Septal Pacing | RV Apical Pacing | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Clinical Event (AT/AF Pnly or Composite of Worsening of Heart Failure, Stroke or Death) Rate From Baseline to Two Year Follow-up
Description: Clinical event (AT/AF pnly or composite of worsening of heart failure, stroke or death) rate from baseline to two year follow-up will be estimated and compared between the group of pacing at RV Mid-Septum and the group of pacing at Apex to identify if pacing at selective RV sites (Mid-Septum or Apex) will have a different long term impact on clinical event rate.
Time Frame: Baseline and 24 months
Population: Data required for the analysis were not collected due to early study termination. Analysis will not be done.
Arm/Group | RV Mid-Septal Pacing | RV Apical Pacing | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Clinical Event (Composite of Worsening of Heart Failure, Stroke or Death) Rate From Baseline to 2 Year Follow-up
Description: Clinical event (composite of worsening of heart failure, stroke or death) rate from baseline to 2 year follow-up will be estimated and compared between the group of pacing at RV Mid-Septum and the group of pacing at Apex to identify if pacing at selective RV sites (Mid-Septum or Apex) will have a different long term impact on clinical event(composite of worsening of heart failure, stroke or death)rate.
Time Frame: Baseline and 24 months
Population: Data required for the analysis were not collected due to early study termination. Analysis will not be done.
Arm/Group | RV Mid-Septal Pacing | RV Apical Pacing | Not Randomized
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events reported before the study termination were included.
Description: Adverse Events were not separated by randomization assignment as there was no subject data analysis completed due to early study termination. All Adverse Events were reviewed by a Central Adverse Event Advisory Committee.
  All serious adverse events were reported. All non-serious adverse events were reported in the table "other adverse events".
Groups:
- Subjects With Implant: All 198 subjects with implant were included in this group.
Arm/Group | Subjects With Implant
Serious Adverse Events (participants affected / at risk) | 50/198
Other Adverse Events (participants affected / at risk) | 12/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Implant (N=198)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 4 (4)
Cardiac perforation (Cardiac disorders) | 5 (5)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Device failure (Injury, poisoning and procedural complications) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Failure to capture (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Lead dislodgement (Injury, poisoning and procedural complications) | 3 (3)
Loss of consciousness (Nervous system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Implant (N=198)
Abdominal mass (Gastrointestinal disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Cardiac flutter (Cardiac disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Lead dislodgement (Injury, poisoning and procedural complications) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pacemaker generated arrhythmia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Early study termination due to enrollment rates significantly below protocol expectations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigational Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication.